CLINICAL TRIAL: NCT03287089
Title: Nitrofurantoin Administration for the Prevention of Short-Term Catheter Associated Urinary Tract Infection After Pelvic Surgery (NAUTICA): A Randomized Controlled Trial
Brief Title: Nitrofurantoin Administration for the Prevention of Short-Term Catheter Associated Urinary Tract Infection After Pelvic Surgery
Acronym: NAUTICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00022622
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2020-05

CONDITIONS: Catheter-Associated Urinary Tract Infection
Keywords: Nitrofurantoin; Prolapse; Pelvic Organ Prolapse; Anti-incontinence procedure; Urinary retention; Urinary Tract Infection; Short-term catheterization
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse; Urinary Retention; Urinary Tract Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitrofurantoin (Active Comparator): Receives twice daily 100mg nitrofurantoin for 5 days following catheter removal
  Interventions: Drug: Nitrofurantoin 100 MG
- Placebo (Placebo Comparator): Receives twice daily matching placebo for 5 days following catheter removal
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Nitrofurantoin 100 MG — Patients will receive nitrofurantoin 100mg twice daily by mouth for 5 days
  Arms: Nitrofurantoin
Drug: Placebo Oral Tablet — Matching placebo
  Arms: Placebo

SUMMARY:
The specific aim of this randomized double-blind placebo-controlled trial is to evaluate the efficacy of administration of nitrofurantoin prophylaxis after catheter discontinuation for the prevention of catheter-associated urinary tract infections in patients with postoperative short-term catheterization following pelvic reconstructive surgery and/or urinary incontinence surgery.

Patients that undergo pelvic organ prolapse and/or urinary incontinence surgery and fail their post-operative voiding trial will be included in the study. Upon successfully passing and in-office voiding trial at the time of catheter removal, they will be randomized to either nitrofurantoin 100mg twice daily or an identical appearing placebo capsule twice daily for 5 days following catheter removal. The primary outcome will be the treatment of clinically suspected and/or culture-proven UTI within 30 days of surgery. Secondary outcomes include adverse events associated with nitrofurantoin use and medication compliance.

Primary and secondary outcomes will be evaluated with Student t test and chi squared or Fisher exact test as appropriate. Assuming a decrease in symptomatic UTIs attributable to nitrofurantoin prophylaxis from 32% to 14%, with 80% power, and a two-sided alpha of 0.05, we should recruit a total of 164 patients.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are the most common hospital-acquired infections, accounting for nearly 30% of cases of nosocomial infections and affecting nearly 1 million people per year.

Following pelvic reconstructive and urinary incontinence surgery, UTIs are one of the most common complications with a risk between 8.9%-34%. The baseline risk of UTI associated with pelvic floor surgery ranges between 5-35%, increasing greatly with catheterization.

Postoperative voiding dysfunction and incomplete bladder emptying is common following pelvic reconstructive and incontinence surgeries, with incidence ranging from 2.5 % to 31%. As a result, these women may have additional catheterization for a short period of time, which increases the risk of UTI. There is a 15-20% risk of developing a postoperative UTI with short-term catheterization, even if the catheter remains in place for merely 24 hours. The risk of UTI increases 5-10% each day the catheter is left in place.

Numerous studies have been conducted to evaluate different prophylactic antibiotic regimens to help decrease the rate of postoperative catheter-associated UTIs. Many of these studies have shown precedent for the use of antibiotic prophylaxis.

Nitrofurantoin has been evaluated as a prophylactic regimen for use during short-term catheterization. These studies had favorable results, decreasing the incidence of UTI postoperatively.

Although there are a few studies showing favorable results for the use of prophylactic nitrofurantoin during catheterization after pelvic surgery, the optimal timing of antibiotic administration and length of dosing regimen is not well defined. The American Urological Association (AUA) recommends empiric antibiotic treatment at the time of external urinary catheter removal in patients with risk factors, such as tobacco use, advanced age, and anatomic abnormalities of the urinary tract. The AUA Panel does cite that bacteriuria in the setting of noninfectious urinary tract disease is a risk factor for bacteremia, and, thus, prophylactic antibiotic treatment at time the of catheter removal may be indicated. The AUA does recommend empiric antibiotic treatment at the removal of an external urinary catheter in patients with risk factors. However, there is no standardization concerning the type of antibiotic to be used or treatment duration.

Although there are a few studies showing favorable results for use of nitrofurantoin during catheterization after pelvic surgery, there are no clearly defined recommendations regarding its use for urinary tract infection prevention after catheter removal. Therefore, the objective of our study is to examine the effects of administration of nitrofurantoin therapy at the time of Foley catheter removal for the prevention of catheter-associated UTI in patients undergoing POP and/or urinary incontinence surgery.

Primary Objective:

To evaluate the efficacy of administration of nitrofurantoin prophylaxis after catheter discontinuation for the prevention of catheter-associated urinary tract infections in patients with postoperative short-term catheterization following pelvic reconstructive surgery. The primary outcome will be the treatment of clinically suspected and/or culture-proven UTI within 30 days of surgery.

Secondary Objective:

To evaluate adverse outcomes related to study medications in each group and to evaluate medication compliance

Null Hypothesis:

The null hypothesis is that the administration of nitrofurantoin will not reduce the rate of UTI compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18
* Creatinine clearance greater than 30 ml/min
* Failed postoperative hospital voiding trial

Exclusion Criteria:

* Pregnant
* History of glucose-6-phosphate dehydrogenase deficiency
* History of renal insufficiency, renal transplant, or nephropathy
* Allergy to nitrofurantoin
* History of recurrent UTI (defined as greater than two culture-proven infections in six months or three infections in one year)
* Urinary Tract Infection (UTI) within 14 days one month of surgery
* Non-English speaking
* Urinary tract infection while Foley catheter is in place
* On antibiotic therapy for other non-urological reasons
* Sustained intraoperative bladder injury requiring prolonged catheterization greater than 5 days
* Undergoing mesh excision from within the bladder, fistula repair, cystotomy repair, urethral diverticulectomy, sacral neuromodulation, urethral surgery, or any other procedure requiring prolonged catheterization and bladder decompression
* Placement of a suprapubic catheter
* Participants that request intermittent self-catheterization
* Neurologic conditions affecting urinary tract system and normal voiding mechanisms
* History of hepatic impairment due to prior nitrofurantoin use
* Inability to provide consent/decisionally impaired
* More than two in-office voiding trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Bastawros, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Wall E, Verkooyen RP, Mintjes-de Groot J, Oostinga J, van Dijk A, Hustinx WN, Verbrugh HA. Prophylactic ciprofloxacin for catheter-associated urinary-tract infection. Lancet. 1992 Apr 18;339(8799):946-51. doi: 10.1016/0140-6736(92)91529-h. PMID 1348797
- [Background] Ghezzi F, Serati M, Cromi A, Uccella S, Salvatore S, Bolis P. Prophylactic single-dose prulifloxacin for catheter-associated urinary tract infection after tension-free vaginal tape procedure. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Jul;18(7):753-7. doi: 10.1007/s00192-006-0233-4. Epub 2006 Nov 21. PMID 17120175
- [Background] Dieter AA, Amundsen CL, Edenfield AL, Kawasaki A, Levin PJ, Visco AG, Siddiqui NY. Oral antibiotics to prevent postoperative urinary tract infection: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):96-103. doi: 10.1097/AOG.0000000000000024. PMID 24463669
- [Background] Jackson D, Higgins E, Bracken J, Yandell PM, Shull B, Foster RT Sr. Antibiotic prophylaxis for urinary tract infection after midurethral sling: a randomized controlled trial. Female Pelvic Med Reconstr Surg. 2013 May-Jun;19(3):137-41. doi: 10.1097/SPV.0b013e318285ba53. PMID 23611930
- [Background] Sutkin G, Alperin M, Meyn L, Wiesenfeld HC, Ellison R, Zyczynski HM. Symptomatic urinary tract infections after surgery for prolapse and/or incontinence. Int Urogynecol J. 2010 Aug;21(8):955-61. doi: 10.1007/s00192-010-1137-x. Epub 2010 Mar 31. PMID 20354678
- [Background] Dieter AA, Amundsen CL, Visco AG, Siddiqui NY. Treatment for urinary tract infection after midurethral sling: a retrospective study comparing patients who receive short-term postoperative catheterization and patients who pass a void trial on the day of surgery. Female Pelvic Med Reconstr Surg. 2012 May-Jun;18(3):175-8. doi: 10.1097/SPV.0b013e3182544e03. PMID 22543772
- [Background] Vigil HR, Mallick R, Nitti VW, Lavallee LT, Breau RH, Hickling DR. Risk Factors for Urinary Tract Infection following Mid Urethral Sling Surgery. J Urol. 2017 May;197(5):1268-1273. doi: 10.1016/j.juro.2016.12.093. Epub 2016 Dec 27. PMID 28034608
- [Background] Schiotz HA, Guttu K. Value of urinary prophylaxis with methenamine in gynecologic surgery. Acta Obstet Gynecol Scand. 2002 Aug;81(8):743-6. doi: 10.1080/j.1600-0412.2002.810810.x. PMID 12174159
- [Background] Albo ME, Richter HE, Brubaker L, Norton P, Kraus SR, Zimmern PE, Chai TC, Zyczynski H, Diokno AC, Tennstedt S, Nager C, Lloyd LK, FitzGerald M, Lemack GE, Johnson HW, Leng W, Mallett V, Stoddard AM, Menefee S, Varner RE, Kenton K, Moalli P, Sirls L, Dandreo KJ, Kusek JW, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Burch colposuspension versus fascial sling to reduce urinary stress incontinence. N Engl J Med. 2007 May 24;356(21):2143-55. doi: 10.1056/NEJMoa070416. Epub 2007 May 21. PMID 17517855
- [Background] Sutkin G, Lowder JL, Smith KJ. Prophylactic antibiotics to prevent urinary tract infection during clean intermittent self-catheterization (CISC) for management of voiding dysfunction after prolapse and incontinence surgery: a decision analysis. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Aug;20(8):933-8. doi: 10.1007/s00192-009-0885-y. Epub 2009 Apr 10. PMID 19582384
- [Background] Falagas ME, Athanasiou S, Iavazzo C, Tokas T, Antsaklis A. Urinary tract infections after pelvic floor gynecological surgery: prevalence and effect of antimicrobial prophylaxis. A systematic review. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1165-72. doi: 10.1007/s00192-008-0584-0. Epub 2008 Apr 10. PMID 18401538
- [Background] Rogers RG, Kammerer-Doak D, Olsen A, Thompson PK, Walters MD, Lukacz ES, Qualls C. A randomized, double-blind, placebo-controlled comparison of the effect of nitrofurantoin monohydrate macrocrystals on the development of urinary tract infections after surgery for pelvic organ prolapse and/or stress urinary incontinence with suprapubic catheterization. Am J Obstet Gynecol. 2004 Jul;191(1):182-7. doi: 10.1016/j.ajog.2004.03.088. PMID 15295362
- [Background] Wolf SJ, Bennett CJ, Dmochowski RR et al. (2012). Urologic Surgery Antimicrobial Prophylaxis. American Urological Association. Retrieved from http://www.auanet.org/guidelines/antimicrobial-prophylaxis-(2008-reviewed-and-validity-confirmed-2011-amended-2012)
- [Background] Harding GK, Nicolle LE, Ronald AR, Preiksaitis JK, Forward KR, Low DE, Cheang M. How long should catheter-acquired urinary tract infection in women be treated? A randomized controlled study. Ann Intern Med. 1991 May 1;114(9):713-9. doi: 10.7326/0003-4819-114-9-713. PMID 2012351
- [Background] Niel-Weise BS, van den Broek PJ. Antibiotic policies for short-term catheter bladder drainage in adults. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD005428. doi: 10.1002/14651858.CD005428. PMID 16034973
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Rodriguez-Martinez JM, Ballesta S, Pascual A. Activity and penetration of fosfomycin, ciprofloxacin, amoxicillin/clavulanic acid and co-trimoxazole in Escherichia coli and Pseudomonas aeruginosa biofilms. Int J Antimicrob Agents. 2007 Oct;30(4):366-8. doi: 10.1016/j.ijantimicag.2007.05.005. Epub 2007 Jul 5. No abstract available. PMID 17616359
- [Background] Sastry S, Doi Y. Fosfomycin: Resurgence of an old companion. J Infect Chemother. 2016 May;22(5):273-80. doi: 10.1016/j.jiac.2016.01.010. Epub 2016 Feb 28. PMID 26923259
- [Background] Jancel T, Dudas V. Management of uncomplicated urinary tract infections. West J Med. 2002 Jan;176(1):51-5. doi: 10.1136/ewjm.176.1.51. No abstract available. PMID 11788540
- [Background] Goettsch WG, Janknegt R, Herings RM. Increased treatment failure after 3-days' courses of nitrofurantoin and trimethoprim for urinary tract infections in women: a population-based retrospective cohort study using the PHARMO database. Br J Clin Pharmacol. 2004 Aug;58(2):184-9. doi: 10.1111/j.1365-2125.2004.02106.x. PMID 15255801
- [Derived] Bastawros D, Kaczmarski K, Zhao J, Bender R, Myers E, Tarr ME. Twice-Daily Nitrofurantoin Administration Following Short-term Transurethral Catheterization After Pelvic Reconstructive Surgery: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Mar 1;27(3):202-207. doi: 10.1097/SPV.0000000000000977. PMID 33620905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive women were prescreened for eligibility and introduced to the study prior to surgery. Women with postoperative urinary retention following pelvic organ prolapse and/or incontinence surgery were approached for study inclusion at the time of their postoperative in-office voiding trial between September 2017 and April 2019.
Pre-assignment Details: Women were deemed as "enrolled" once they consented and randomized. No enrolled participants were excluded with this definition.
Period: Overall Study
Arm/Group | Nitrofurantoin | Placebo
Started | 82 | 82
Completed | 82 | 76
Not Completed | 0 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analyses were conducted on Intention-to-Treat Principle
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrofurantoin | Placebo | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.7) | 61.1 (12.4) | 61.4 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 82 | 82 | 164
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 79 | 72 | 151
  Black | 1 | 8 | 9
  Other | 2 | 2 | 4
Body Mass Index (BMI), kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.7) | 28.6 (5) | 27.8 (4.9)
Parity [Median (Inter-Quartile Range); unit: Parity] | 2 [1 to 3] | 2 [2 to 3] | 2 [2 to 3]
POP-Q Stage [Median (Inter-Quartile Range); unit: units on a scale] — POP-Q is a measure of the degree of Pelvic Organ Prolapse present. Stage 0 is essentially no prolapse or descent of pelvic organs; higher stages indicate progressively larger degrees of prolapse. Stage 4 is the highest stage, and indicated prolapse that is equal to or greater than the total vaginal length (in cm) minus 2 cm
  units on a scale | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 18 | 17 | 35
  Postmenopausal | 64 | 64 | 128
  Missing data | 0 | 1 | 1
Postmenopausal Hormone Use [Count of Participants; unit: Participants]
  No Hormone Therapy | 58 | 58 | 116
  Vaginal Estrogen Therapy | 20 | 19 | 39
  Systemic Hormonal Therapy | 4 | 5 | 9
Current Smoking [Count of Participants; unit: Participants] | 6 | 6 | 12
History of Recurrent UTI [Count of Participants; unit: Participants] | 1 | 1 | 2
Diabetes Mellitus [Count of Participants; unit: Participants] | 9 | 10 | 19
Preoperative PVR Volume (mL) [Mean (Standard Deviation); unit: mL] | 57.9 (92.6) | 45.3 (55.7) | 51.4 (75.5)
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min] | 84.1 (30.1) | 94.2 (34.9) | 89.1 (32.9)
Type of Procedure [Count of Participants; unit: Participants] — Participants may have had more than one procedure listed
  Participants
    Mid urethral sling surgery | 50 | 47 | 97
    Burch colposuspension | 1 | 2 | 3
    Anterior repair | 15 | 20 | 35
    Posterior repair | 53 | 59 | 112
    Hysterectomy | 32 | 35 | 67
    Vaginectomy/colpocleisis | 7 | 2 | 9
    Uterosacral ligament suspension | 18 | 24 | 42
    Sacrospinous ligament fixation | 0 | 1 | 1
    Iliococcygeus vault suspension | 1 | 1 | 2
    Sacral colpopexy | 4 | 1 | 5
    Vaginal mesh excision | 4 | 1 | 5
Operative Time (mins) [Mean (Standard Deviation); unit: minutes] | 134 (80.8) | 142.9 (86.9) | 138.4 (83.8)
Estimated Blood Loss (mL) [Mean (Standard Deviation); unit: mL] | 45.5 (35.5) | 60.9 (61.6) | 53.2 (50.7)
Length of Hospital Stay (days) [Median (Inter-Quartile Range); unit: days] | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]
Duration of Catheterization (days) [Median (Inter-Quartile Range); unit: days] | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: UTI
Description: Number of participants with a urinary tract infection in the first 30 days following pelvic reconstructive surgery
Time Frame: within 30 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 82 | 82
Participants | 15 | 14
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 0.84, Chi-squared; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.49 to 2.43]

2. Secondary Outcome: Adverse Events
Description: Number of participants with an adverse event only related to study drug administration
Time Frame: within 30 days of surgery
Population: This is the total number of participants with an allergy or intolerance to the study medication.These adverse symptoms included: hives, pruritus, rash, anaphylaxis, nausea, vomiting, diarrhea, and other.
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 5 | 4
Participants
  Allergy | 0 | 0
  Nausea | 5 | 2
  Vomiting | 0 | 0
  Diarrhea | 0 | 0
  Other | 0 | 2
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 0.44, Chi-squared

3. Secondary Outcome: Medication Compliance
Description: Compliance assessed by use of a medication diary during treatment period
Time Frame: within 30 days of surgery
Population: Compliance was defined as the number pills taken divided by total number of pills dispensed (10). The closer this ratio is to "1" the better the compliance. The closer the ratio is to "0" the worse the compliance
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 82 | 82
ratio | 0.95 (0.18) | 0.96 (0.15)
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 0.68, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 30 days (from surgery until 30 days postop)
Description: Adverse events data related to study medication was collected (i.e. allergies and/or intolerances)
Arm/Group | Nitrofurantoin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 5/82 | 4/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrofurantoin (N=82) | Placebo (N=82)
Medication Intolerance (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Joint Pain
Medication Intolerance (Gastrointestinal disorders) | 5 (5) | 2 (2) — Nausea
Medication Intolerance (General disorders) | 0 (0) | 1 (1) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03287089/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03287089/ICF_001.pdf